CLINICAL TRIAL: NCT01922076
Title: A Phase 1 Study of AZD1775 (MK-1775) Concurrent With Local Radiation Therapy for the Treatment of Newly Diagnosed Children With Diffuse Intrinsic Pontine Gliomas
Brief Title: Adavosertib and Local Radiation Therapy in Treating Children With Newly Diagnosed Diffuse Intrinsic Pontine Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01602; NCI-2013-01602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL1217; ADVL1217 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1217 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligoastrocytoma; Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma, H3 K27M-Mutant; Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Astrocytoma; Diffuse Intrinsic Pontine Glioma; Glioblastoma; Gliosarcoma | interventions — adavosertib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (adavosertib, radiation therapy) (Experimental): Patients undergo radiation therapy 5 days a week for 6 weeks (up to 30 fractions). Patients also receive adavosertib PO on days 1-5 of weeks 1, 3, and 5; days 1-5 of weeks 1, 3, and 5 AND days 1, 3, and 5 of weeks 2, 4, and 6; OR days 1-5 of weeks 1-6 depending on dose level assignment. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects and the best dose of adavosertib when given together with local radiation therapy in treating children with newly diagnosed diffuse intrinsic pontine gliomas. Adavosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays, gamma rays, neutrons, protons, or other sources to kill tumor cells and shrink tumors. Giving adavosertib with local radiation therapy may work better than local radiation therapy alone in treating diffuse intrinsic pontine gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) or recommended phase 2 dose and schedule of the adavosertib (Wee1 inhibitor AZD1775 [MK-1775]) administered concurrently with radiation therapy in children with newly diagnosed diffuse intrinsic pontine glioma (DIPG).

II. To define and describe the toxicities of AZD1775 (MK-1775) given concurrently with radiation therapy in children with newly diagnosed DIPG.

III. To characterize the pharmacokinetics of AZD1775 (MK-1775) in children with newly diagnosed DIPG when given concurrently with radiation therapy.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of AZD1775 (MK-1775) within the confines of a phase 1 study, including response rate, progression free survival, and overall survival of treated patients.

II. To assess the biologic activity of AZD1775 (MK-1775) by measuring expression of phosphorylated-cell division cycle 2 G1 to S and G2 to M (p-CDC2) (cyclin-dependent kinase 1 [CDK1]) and phosphorylated-histone H3 (p-HH3) in peripheral blood mononuclear cells (PBMCs) before and after administration of AZD1775 (MK-1775) in children with newly diagnosed DIPG.

III. To assess the biologic activity of AZD1775 (MK-1775) by measuring expression of gamma-H2A histone family, member X (H2AX) in PBMCs, a marker of deoxyribonucleic acid (DNA) double-strand breaks (dsDNA), before and after administration of AZD1775 (MK-1775) in children with newly diagnosed DIPG.

OUTLINE: This is a dose-escalation study of adavosertib.

Patients undergo radiation therapy 5 days a week for 6 weeks (up to 30 fractions). Patients also receive adavosertib orally (PO) on days 1-5 of weeks 1, 3, and 5; days 1-5 of weeks 1, 3, and 5 AND days 1, 3, and 5 of weeks 2, 4, and 6; OR days 1-5 of weeks 1-6 depending on dose level assignment. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 2 months for 6 months, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed DIPGs, defined as tumors with a pontine epicenter and diffuse involvement of the pons, are eligible without histologic confirmation

  * Patients with brainstem tumors that do not meet these criteria or are not considered to be typical intrinsic pontine gliomas will only be eligible if the tumors are biopsied and proven to be an anaplastic astrocytoma, glioblastoma, gliosarcoma, diffuse midline glioma with histone H3 K27M mutation, or anaplastic mixed glioma; patients with pilocytic astrocytoma, fibrillary astrocytoma, gangliogliomas, or other mixed gliomas without anaplasia are not eligible
  * Patients with disseminated disease are not eligible, and magnetic resonance imaging (MRI) of spine must be performed if disseminated disease is suspected by the treating physician
  * Enrollment must be no later than 28 days after the date of radiographic diagnosis or surgery, whichever is the later date
* Patients must have a body surface area >= 0.35 m^2 at the time of study enrollment
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must not have received any prior anti-cancer therapy such as chemotherapy, radiation therapy, immunotherapy or bone marrow transplant for the treatment of DIPG; prior dexamethasone and/or surgery are allowed
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or
* A serum creatinine based on age/gender as follows:

  * 0.8 mg/dL (3 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dl (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dl (female) (>= 16 years of age)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN = 135 units per liter (U/L); for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum glutamic oxaloacetic transaminase (SGOT) aspartate aminotransferase [AST] =< 3 x ULN = 150 U/L; for the purpose of this study, the ULN for SGOT is 50 U/L
* Serum albumin >= 2 g/dL
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v]5) resulting from prior therapy must be =< grade 2 with the exception of tendon reflex (deep tendon reflex [DTR]); any grade of DTR is eligible
* Corrected QT interval (QTc) =< 480 msec
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women may not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; negative serum or urine pregnancy test within 3 days prior to enrollment
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive methods as follows: fertile females of childbearing potential who agree to use adequate contraceptive measures from 2 weeks prior to the study and until 1 month after study treatment discontinuation; male patients willing to abstain or use barrier contraception (i.e. condoms) for the duration of the study and for 3 months after treatment stops
* Patients receiving corticosteroids are eligible for this trial
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients must not currently be receiving enzyme inducing anticonvulsants
* Patients should avoid concomitant medication known or suspected to prolong QTc interval or cause Torsades De Pointes; if possible, alternative agents should be considered; patients who are receiving drugs that prolong the QTc are eligible if the drug is necessary and no alternatives are available
* Patients who are currently receiving drugs that are strong or moderate inhibitors and/or inducers of CYP3A4, sensitive CYP3A4 substrates and CYP3A4 substrates with a narrow therapeutic range are not eligible; the use of aprepitant or fosaprepitant as an antiemetic is prohibited due to early drug interaction data demonstrating increased exposure to AZD1775; the use of hydroxymethylglutary (HMG) coenzyme-A (Co-A) inhibitors such as atorvastatin is prohibited
* Herbal preparations are not allowed throughout the study; these herbal medications include but are not limited to: St. John's wort, kava, ephedra (ma hung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto and ginseng; patients should stop using these herbal medications 7 days prior to study enrollment
* Any known hypersensitivity or contraindication to the components of the study drug AZD1775
* Patients must not receive metformin for at least 5 days prior to enrollment and for the duration of study treatment
* Patients must be able to swallow capsules; nasogastric or gastrostomy feeding (G) tube administration is not allowed
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients with cardiac diseases ongoing or in the past 6 months (e.g. congestive heart failure, acute myocardial infarction, significant uncontrolled arrhythmias) are not eligible for this trial
* Major surgical procedures =< 28 days of beginning study treatment, or minor surgical procedures (including ventriculoperitoneal [VP] shunt placement or stereotactic biopsy of the tumor) =< 7 days; no waiting period required following port-a-cath or other central venous access placement
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 37 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mueller, Principal Investigator — COG Phase I Consortium
Locations (24):
- United States (23):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 50 mg/m^2: Patients receive 50 mg/m^2 adavosertib daily (Monday- Friday), alternating weeks.
- Dose Level 2: 50 mg/m^2: Patients receive 50 mg/m^2 adavosertib daily (Monday-Friday), alternating with weeks of QOD dosing.
- Dose Level 3: 50 mg/m^2: Patients receive 50 mg/m^2 adavosertib daily (Monday- Friday), during weeks 1-6
- Dose Level 4: 95 mg/m^2: Patients receive 95 mg/m^2 adavosertib daily (Monday- Friday), during weeks 1-6
- Dose Level 5: 130 mg/m^2: Patients receive 130 mg/m^2 adavosertib daily (Monday- Friday), during weeks 1-6
- Dose Level 6: 160 mg/m^2: Patients receive 160 mg/m^2 adavosertib daily (Monday- Friday), during weeks 1-6
- Dose Level 7: 200 mg/m^2: Patients receive 200 mg/m^2 adavosertib daily (Monday- Friday), during weeks 1-6
Period: Overall Study
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Started | 6 | 6 | 7 | 7 | 7 | 6 | 7
Completed | 6 | 6 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 1 | 1 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2 | Total
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 7 | 7 | 7 | 5 | 7 | 45
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 8 [6.0 to 18.0] | 5.5 [3.0 to 9.0] | 6 [3.0 to 8.0] | 6 [4.0 to 8.0] | 6 [5.0 to 12.0] | 5.5 [3.0 to 21.0] | 7 [3.0 to 13.0] | 6 [3.0 to 21.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 4 | 5 | 4 | 4 | 24
  Male | 5 | 3 | 4 | 3 | 2 | 2 | 3 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 3 | 0 | 1 | 1 | 7
  Not Hispanic or Latino | 5 | 6 | 6 | 4 | 7 | 5 | 6 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 6
  White | 5 | 4 | 5 | 3 | 5 | 2 | 4 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 1 | 0 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose of Adavosertib
Description: MTD will be defined as the maximum dose at which fewer than one-third of patients experience a dose-limiting toxicity graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 42 days
Population: All eligible patients
Measure: Number; unit: mg/m^2
Groups:
- Treatment (Adavosertib): Patients also receive adavosertib PO on days 1-5 of weeks 1, 3, and 5; days 1-5 of weeks 1, 3, and 5 AND days 1, 3, and 5 of weeks 2, 4, and 6; OR days 1-5 of weeks 1-6 depending on dose level assignment. Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Adavosertib)
Number analyzed (Participants) | 46
mg/m^2 | 200

2. Primary Outcome: Number of Dose Limiting Toxicity With Adavosertib
Description: Number of patients with dose limiting toxicity stratified by dose level and the toxicity will be graded using the NCI CTCAE version 4.0.
Time Frame: Up to 42 days
Population: All Toxicity evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 5 | 6
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 1

3. Primary Outcome: Area Under the Time Concentration Curve of Adavosertib
Description: Median (min, max) of the area under the concentration time curve adavosertib assessed at 1, 2, 4, 6, 8, and 24 hours post dose on day 1 stratified by dose level and study part.
Time Frame: up to 24 hours
Population: All eligible patients
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7
hr*ng/mL | 1122.2 [918.1 to 1839.4] | 1233.3 [540.5 to 1511.7] | 777.3 [394.1 to 1346.3] | 2863.5 [1503.2 to 3692.4] | 2525.5 [1650.5 to 4547.6] | 5996.2 [3413.7 to 7042.9] | 5781.6 [5007.2 to 6556.0]

4. Secondary Outcome: Number of Patients With Response to Adavosertib
Description: Number of participants with response (CR/PR) by maximal 2-dimensional measures with CR: disappearance of all abnormal signal within the brainstem; PR: at least 50% decrease in the sum o the products of the two perpendicular diameters of the target lesion.
Time Frame: Up to 4 years
Population: All response evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 7 | 5 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS) of Adavosertib
Description: Median (95% CI) time to progression or death stratified by dose level and study part. PFS was defined as time from start date of the first treatment to the date of disease progression or death due to any causes which ever occurred first.
Time Frame: Up to 4 years
Population: All response evaluable patients
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 7 | 5 | 6
Days | 426.5 [233 to 521] | 250 [229 to 421] | 450.5 [307 to 497] | 333 [189 to 394] | 260 [209 to 558] | 264 [72 to 1032] | 406 [300 to 753]

6. Secondary Outcome: Overall Survival (OS) of Adavosertib
Description: Median (95% CI) time to progression or death stratified by dose level and study part.
Time Frame: Up to 4 years
Population: All response evaluable patients
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 7 | 5 | 6
Days | 426.5 [312 to 521] | 250 [229 to 421] | 450.5 [307 to 497] | 372.5 [272 to 560] | 274 [219 to 558] | 273 [72 to NA] — The upper limit of the 95% CI is not estimable because the upper limit of the 95% confidence bands does not reach 0.50. This occurs in instances when not enough events have occurred to estimate the parameter. | 406 [300 to 752]

7. Secondary Outcome: Change in p-CDC2 of Adavosertib
Description: Median (min, max) change in expression of p-CDC2 in peripheral blood mononuclear cells (PBMCs) before and after administration by dose level and study part.
Time Frame: Baseline to day 8
Population: Data were not and will never be collected.
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Change in Expression of p-HH3 of Adavosertib
Description: Median (min, max) change in expression of p-HH3 in peripheral blood mononuclear cells (PBMCs) before and after administration by dose level and study part
Time Frame: Baseline to day 8
Population: Data were not and will never be collected.
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Change in Expression of ɤ(Gamma)-H2AX of Adavosertib
Description: Median (min, max) relative change in expression of gamma-H2AX of adavosertib by dose level and study part.
Time Frame: Baseline to day 8
Measure: Median (Full Range); unit: ratio
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
ratio | 0.9 [0.6 to 1.6] | 0.9 [0.7 to 1.3] | 0.9 [0.6 to 1.2] | 1.1 [0.2 to 1.8] | 0.9 [0.5 to 1.4] | 1 [0.9 to 1.1] | 1.1 [0.8 to 1.2]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Dose Level 1: 50 mg/m^2 | Dose Level 2: 50 mg/m^2 | Dose Level 3: 50 mg/m^2 | Dose Level 4: 95 mg/m^2 | Dose Level 5: 130 mg/m^2 | Dose Level 6: 160 mg/m^2 | Dose Level 7: 200 mg/m^2
All-Cause Mortality (participants affected / at risk) | 4/6 | 4/6 | 4/7 | 4/7 | 6/7 | 4/6 | 4/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/7 | 2/7 | 2/7 | 2/6 | 1/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 7/7 | 7/7 | 7/7 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: 50 mg/m^2 (N=6) | Dose Level 2: 50 mg/m^2 (N=6) | Dose Level 3: 50 mg/m^2 (N=7) | Dose Level 4: 95 mg/m^2 (N=7) | Dose Level 5: 130 mg/m^2 (N=7) | Dose Level 6: 160 mg/m^2 (N=6) | Dose Level 7: 200 mg/m^2 (N=7)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: 50 mg/m^2 (N=6) | Dose Level 2: 50 mg/m^2 (N=6) | Dose Level 3: 50 mg/m^2 (N=7) | Dose Level 4: 95 mg/m^2 (N=7) | Dose Level 5: 130 mg/m^2 (N=7) | Dose Level 6: 160 mg/m^2 (N=6) | Dose Level 7: 200 mg/m^2 (N=7)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 2 | 2 | 0 | 1 | 0
Abducens nerve disorder (Nervous system disorders) | 4 | 3 | 5 | 3 | 4 | 2 | 3
Accessory nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 3 | 3 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 3 | 2 | 3 | 4 | 4
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 0 | 3 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 3 | 4 | 2 | 5
Anorexia (Metabolism and nutrition disorders) | 5 | 0 | 3 | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0 | 2 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 2 | 1 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 4 | 3 | 4 | 3 | 3 | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood and lymphatic system disorders - Other, EOSINOPHILIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blurred vision (Eye disorders) | 1 | 2 | 2 | 1 | 0 | 1 | 0
Body odor (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac disorders - Other, SYSTOLIC HEART MURMUR (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholesterol high (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 5 | 5 | 4 | 3 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 3 | 2 | 2 | 1
Creatinine increased (Investigations) | 1 | 0 | 2 | 1 | 1 | 1 | 0
Cushingoid (Endocrine disorders) | 3 | 0 | 2 | 2 | 2 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 2 | 1 | 2 | 2 | 3 | 3 | 0
Dysesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 2 | 4 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Edema face (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Edema trunk (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, ANISOCORIA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, DIPLOPIA (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, DOUBLE VISION (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, ESOTROPIA (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, EYE IRRITATION (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, IRRITATION FROM SWIMMING (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, ITCHY EYE (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, LEFT EYELID IRRITATION/ULCERATION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, RIGHT EYELID IRRITATION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, STRABISMUS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, VISION CHANGES (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0
Eyelid function disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 4 | 1 | 4 | 5 | 6 | 1 | 5
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 3 | 3 | 5 | 2 | 2 | 4
Fever (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
GGT increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 2 | 1 | 1 | 3 | 3 | 3 | 3
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, DIFFICULTY CHEWING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
General disorders and administration site conditions - Other, INCREASED APPETITE (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 1
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 | 0 | 2 | 1 | 3 | 0 | 1
Headache (Nervous system disorders) | 4 | 4 | 4 | 4 | 3 | 3 | 5
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hemoglobin increased (Investigations) | 0 | 3 | 1 | 2 | 0 | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 1 | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 2 | 3 | 4
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 4 | 3 | 1 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 2 | 3 | 2 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 3
Hypoglossal nerve disorder (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 4 | 1 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 4 | 3 | 5 | 0 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 1 | 1 | 2 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
INR increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
IVth nerve disorder (Nervous system disorders) | 2 | 0 | 1 | 0 | 2 | 1 | 0
Infections and infestations - Other, CANDIDIASIS-ORAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other, ORAL THRUSH (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Infections and infestations - Other, STREP THROAT (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 0 | 2 | 0 | 0 | 1 | 2
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, BILIRUBIN (TOTAL) DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, CHLORIDE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, ANION GAP (ALB CORRECTED) INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, BICARBONATE (TOTAL CO2) DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, BICARBONATE SERUM LOW (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, BLOOD UREA NITROGEN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, CREATININE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, ELEVATED BUN (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Investigations - Other, ELEVATED LDH (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, ELEVTAED BUN (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, LYMPHOCYTE % DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, MEAN CORPUSCULAR HEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, MEAN PLATELET VOLUME DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, MONOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, NEUTROPHIL % INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, PROTEIN (TOTAL) DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 3 | 2 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localized edema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 6 | 6 | 7 | 6 | 5 | 5 | 6
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, HYPERPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Metabolism and nutrition disorders - Other, HYPOPROTEINEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Metabolism and nutrition disorders - Other, INCREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, LOW BICARBONATE, RELATED TO CENTRAL HYPERVENTILATION SYN (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolism and nutrition disorders - Other, POLYPHAGIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 2 | 1 | 2
Muscle weakness left-sided (Nervous system disorders) | 2 | 0 | 1 | 1 | 2 | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 2 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0 | 1 | 1 | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, BILATERAL SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, HYPPEREFLEXIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, JAW PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Mild tenderness with palpation of his oblique muscles and anterior iliac crest.
Musculoskeletal and connective tissue disorder - Other, TWITCHING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 3 | 2 | 3 | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, DISEASE PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 4 | 3 | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Tumor Progresiion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, CENTRAL HYPERVENTILATION SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other, CLONUS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, CONCUSSION (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, DIPLOPIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, DYSDIADOCHOKINESIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, DYSMETRIA (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, HEAD TILT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, HYPERREFLEXIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other, HYPOREFLEXIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, INTERMITTENT HEAD TILT (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, INTRA-TUMORAL HEMORRHAGE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, LEFT TONGUE DEVIATION (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, LUE AND LLE, ALTERED SENSATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other, NYSTAGMUS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorders - Other, SLOWED RESPONSES/REACTIONS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 1 | 0 | 2 | 2 | 5
Nystagmus (Nervous system disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 2
Oculomotor nerve disorder (Nervous system disorders) | 2 | 2 | 2 | 0 | 2 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Papilledema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 | 3 | 2 | 2 | 3 | 3 | 6
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, VIVID DREAMS (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, DIFFICULTY STARTING TO VOID (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, GLUCOSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, KETONURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, URINARY HESITATION (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, URINARY HESTIANCY (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, BRADYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, DECREASED BREATH SOUNDS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, INCREASED WORK OF BREATHING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, PARANASAL SINUS DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 2 | 3 | 1 | 1 | 1
Skin and subcutaneous tissue disorders - Other, ABRASION TO LEFT FOREARM (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, CONTACT DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, DERMATITIS IN AXILLA/ON ABDOMEN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, MOTTLED SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vagus nerve disorder (Nervous system disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2 | 5 | 2 | 3 | 4 | 3
Weight gain (Investigations) | 1 | 1 | 2 | 3 | 0 | 1 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
White blood cell decreased (Investigations) | 5 | 5 | 5 | 4 | 3 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT01922076/Prot_SAP_001.pdf